CLINICAL TRIAL: NCT00300885
Title: A Randomized Controlled Trial Comparing Safety and Efficacy of Carboplatin and Paclitaxel Plus or Minus Sorafenib (BAY 43-9006) in Chemonaive Patients With Stage IIIB-IV Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on the results of the interim analysis, it was determined that the study would not meet its primary efficacy endpoint and the study was terminated early.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11961; 2005-005245-19 (EudraCT Number)
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Results first posted 2010-09-20 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: Non-Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorafenib + C/P (Experimental): Chemotherapy Phase up to 6 cycles: Sorafenib (Nexavar, BAY43-9006), [400 mg orally, twice daily] on Study Days 2-19 and paclitaxel (P) (200 mg/m2, intravenous (IV)) and carboplatin (C) (area under the curve (AUC) =6 mg/ml*min-1, IV) on Study Day 1. The cycle duration 21 days. Maintenance Phase: Sorafenib 400 mg orally twice daily was administered on Days 1-21 of each 21-day cycle.
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006) + carboplatin + paclitaxel
- Placebo + C/P (Active Comparator): Chemotherapy Phase up to 6 cycles: Sorafenib Placebo (2 tablets orally twice daily] on Study Days 2-19 and paclitaxel (200 mg/m2, intravenous (IV)) and carboplatin (area under the curve (AUC) =6 mg/ml*min-1, IV) on Study Day 1. The cycle duration 21 days. Maintenance Phase: Sorafenib Placebo 2 tablets orally twice daily was administered on Days 1-21 of each 21-day cycle.
  Interventions: Drug: Carboplatin plus Paclitaxel

INTERVENTIONS:
Drug: Nexavar (Sorafenib, BAY43-9006) + carboplatin + paclitaxel — Chemotherapy Phase up to 6 cycles: Sorafenib (Nexavar, BAY43-9006), [400 mg orally, twice daily] on Study Days 2-19 and paclitaxel (P) (200 mg/m2, intravenous (IV)) and carboplatin (C) (area under the curve (AUC) =6 mg/ml*min-1, IV) on Study Day 1. The cycle duration 21 days. Maintenance Phase: Sorafenib 400 mg orally twice daily was administered on Days 1-21 of each 21-day cycle.
  Arms: Sorafenib + C/P
Drug: Carboplatin plus Paclitaxel — Chemotherapy Phase up to 6 cycles: Sorafenib Placebo (2 tablets orally twice daily] on Study Days 2-19 and paclitaxel (200 mg/m2, intravenous (IV)) and carboplatin (area under the curve (AUC) =6 mg/ml*min-1, IV) on Study Day 1. The cycle duration 21 days. Maintenance Phase: Sorafenib Placebo 2 tablets orally twice daily was administered on Days 1-21 of each 21-day cycle.
  Arms: Placebo + C/P

SUMMARY:
A randomized controlled trial comparing safety and efficacy of carboplatin and paclitaxel plus or minus sorafenib in chemonaive patients with stage III-IV non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB (with effusion) or Stage IV NSCLC any histology
* No prior chemotherapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Greater than or equal to 18 years of age
* Life expectancy at least 12 weeks
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Prior systemic anti cancer therapy
* Known brain metastasis. Patients with neurological symptoms should undergo at computed tomography (CT) scan/magnetic resonance imaging (MRI) of the brain to exclude brain metastasis
* Pulmonary hemorrhage/bleeding event > Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 within 4 weeks of first dose of study drug
* Thrombotic or embolic events including Transient ischemic attack (TIA) within the past 6 months
* Uncontrolled hypertension
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Major surgery within 4 weeks
* Evidence or history of bleeding diathesis or coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 926 (Actual)
Dates: Start 2006-02; Primary Completion 2007-10 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (180):
- United States (72):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Springdale, Arkansas
  - Anaheim, California
  - Beverly Hills, California
  - Burbank, California
  - Corona, California
  - Encinitas, California
  - Highland, California
  - Los Angeles, California
  - Orange, California
  - Sacramento, California
  - Denver, Colorado
  - Lakeland, Florida
  - Merritt Island, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Skokie, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Kokomo, Indiana
  - Sioux City, Iowa
  - Hutchinson, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Metairie, Louisiana
  - Boston, Massachusetts
  - Pittsfield, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Hattiesburg, Mississippi
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Hackensack, New Jersey
  - Morristown, New Jersey
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Columbus, Ohio
  - Dayton, Ohio
  - Dover, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pottsville, Pennsylvania
  - Sayre, Pennsylvania
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Trophy Club, Texas
  - Salt Lake City, Utah
  - Abingdon, Virginia
  - Fairfax, Virginia
  - Richlands, Virginia
  - Richmond, Virginia
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Argentina (7):
  - El Palomar - Morón, Buenos Aires
  - La Plata, Buenos Aires
  - Mar del Plata, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Rosario, Santa Fe Province
  - Capital Federal-Buenos Aires
  - Santa Fé
- Australia (7):
  - Port Macquarie, New South Wales
  - Wollongong, New South Wales
  - Brisbane, Queensland
  - Adelaide, South Australia
  - Frankston, Victoria
  - Melbourne, Victoria
  - Perth, Western Australia
- Belgium (4):
  - Bruxelles - Brussel
  - Charleroi
  - La Louvière
  - Liège
- Brazil (15):
  - Fortaleza, Ceará
  - Salvador, Estado de Bahia
  - Brasília, Federal District
  - Goiânia, Goiás
  - Nova Lima, Minas Gerais
  - Curitiba, Paraná
  - Porto Alegre, Rio Grande do Sul
  - Joinville, Santa Catarina
  - Barretos, São Paulo
  - Jaú, São Paulo
  - Ribeirão Preto, São Paulo
  - Santo André, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo
  - Belo Horizonte
- Canada (5):
  - North Vancouver, British Columbia
  - Barrie, Ontario
  - Brampton, Ontario
  - Montreal, Quebec
  - Regina, Saskatchewan
- Chile (2):
  - Santiago, Santiago Metropolitan
  - Santiago
- France (7):
  - Bobigny
  - Caen
  - Clamart
  - Metz
  - Nancy
  - Nice
  - Strasbourg
- Germany (15):
  - Heidelberg, Baden-Wurttemberg
  - Mannheim, Baden-Wurttemberg
  - Gauting, Bavaria
  - München, Bavaria
  - Hamburg, Hamburg
  - Hofheim, Hesse
  - Göttingen, Lower Saxony
  - Hanover, Lower Saxony
  - Oldenburg, Lower Saxony
  - Essen, North Rhine-Westphalia
  - Hemer, North Rhine-Westphalia
  - Leverkusen, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Großhansdorf, Schleswig-Holstein
  - Berlin, State of Berlin
- Hong Kong, Hong Kong
- Hungary (5):
  - Budapest
  - Deszk
  - Gyula
  - Mátraháza
  - Törökbálint
- Italy (9):
  - Orbassano, Torino
  - Bergamo
  - Genova
  - Milan
  - Parma
  - Pavia
  - Perugia
  - Roma
  - Torino
- Netherlands (2):
  - Eindhoven, North Brabant
  - Zwolle
- Poland (6):
  - Gdansk
  - Krakow
  - Olsztyn
  - Otwock
  - Warsaw
  - Wroclaw
- San Juan, Puerto Rico
- Russia (2):
  - Moscow
  - Saint Petersburg
- Seoul, South Korea
- Spain (8):
  - Alicante, Alicante
  - Elche, Alicante
  - Zaragoza, Aragon
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Majadahonda, Madrid
  - Pontevedra, Pontevedra
  - Zamora, Zamora
- Sweden (3):
  - Gävle
  - Stockholm
  - Uppsala
- Taiwan (3):
  - Taichung
  - Taipei
  - Taoyuan District
- United Kingdom (5):
  - Plymouth, Devon
  - Bornemouth, Dorset
  - Leicester, Leicestershire
  - London, London
  - Manchester, Manchester

REFERENCES:
- [Result] Scagliotti G, Novello S, von Pawel J, Reck M, Pereira JR, Thomas M, Abrao Miziara JE, Balint B, De Marinis F, Keller A, Aren O, Csollak M, Albert I, Barrios CH, Grossi F, Krzakowski M, Cupit L, Cihon F, Dimatteo S, Hanna N. Phase III study of carboplatin and paclitaxel alone or with sorafenib in advanced non-small-cell lung cancer. J Clin Oncol. 2010 Apr 10;28(11):1835-42. doi: 10.1200/JCO.2009.26.1321. Epub 2010 Mar 8. PMID 20212250
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 150 centers across 20 countries, which enrolled and randomized at least one subject. From a total of 1043 subjects who were screened, 926 subjects were randomized between 15 February 2006 and 9 May 2007 in 20 countries.
Pre-assignment Details: Of the 926 subjects who were randomized, 922 received at least one dose of study drug. All 926 subjects were included in the ITT population (intent-to-treat; defined as all randomized patients), all but four subjects did receive study drug. They were not included in the safety population.
Period: Treatment
Arm/Group | Sorafenib + C/P | Placebo + C/P
Started | 464 | 462 (ongoing in double -blind treatment at data cut-off)
Received Treatment | 463 | 459
Completed | 91 | 88
Not Completed | 373 | 374
Not completed — Adverse Event | 134 | 82
Not completed — Death | 20 | 7
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 4 | 5
Not completed — Protocol Violation | 11 | 11
Not completed — Withdrawal by Subject | 26 | 23
Not completed — Disease progression | 171 | 238
Not completed — Random code broken (subject died) | 0 | 1
Not completed — Non-compliant with study medication | 3 | 4
Period: Follow-up
Arm/Group | Sorafenib + C/P | Placebo + C/P
Started | 354 (Subjects entered Follow-up period after termination of Treatment period due to any reason.) | 369 (Subjects entered Follow-up period after termination of Treatment period due to any reason.)
Completed | 176 (Subjects still in Follow up period at data cut-off date.) | 174 (Subjects still in Follow up period at data cut-off date.)
Not Completed | 178 | 195
Not completed — Death | 141 | 163
Not completed — Lost to Follow-up | 11 | 7
Not completed — Withdrawal by Subject | 26 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib + C/P | Placebo + C/P | Total
Number analyzed (Participants) | 464 | 462 | 926
Age, Continuous [Median (Full Range); unit: years] | 62 [34 to 86] | 63 [34 to 82] | 62 [34 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 174 | 345
  Male | 293 | 288 | 581
ECOG (Eastern Cooperative Oncology Group) Performance Status [Number; unit: Participants] — ECOG 0 versus 1 was a stratification factor for randomization. ECOG Performance Status is a rating of daily living abilities, from 0 to 5: 0= fully active without restriction. 1= restricted in physically strenuous activity; 2= ambulatory, capable of all selfcare; 3= capable of limited selfcare; 4= completely disabled; 5= dead.
  Participants
    0 | 190 | 188 | 378
    1 | 274 | 274 | 548
Geographic region [Number; unit: Participants] — Geographic region (core versus non-core) was stratification factor for randomization. Core region comprises North America, Northern/Western Europe, and Australia. Non-core region comprises South America, Eastern Europe, and Asia-Pacific.
  Participants
    core | 325 | 323 | 648
    non-core | 139 | 139 | 278
NSCLC Classification [Number; unit: Participants] — Histology (squamous versus non-squamous) was a stratification factor for randomization.
  Participants
    Adenocarcinoma NSCLC | 263 | 271 | 534
    Bronchoalveolar | 6 | 5 | 11
    Non-Microcellulare carcinoma | 0 | 1 | 1
    Large cell carcinoma | 23 | 30 | 53
    Squamous cell carcinoma | 109 | 114 | 223
    Non-Small cell lung cancer carcinoma | 10 | 10 | 20
    Undifferentiated carcinoma | 46 | 26 | 72
    Poorly differentiated non-small cell carcinoma | 4 | 3 | 7
    Neuro-Endocrine carcinoma | 0 | 1 | 1
    Low differentiated carcinoma (neuro-endocrine) | 1 | 0 | 1
    Unknown or unspecified histology | 2 | 1 | 3
Stage at Study Entry [Number; unit: Participants] — Stage IIIB (according to American Joint Committee on Cancer): primary tumor any stage, regional lymph node stage N3, no distant metastasis OR primary tumor stage T4, regional lymph node any stage, no distant metastasis. Stage IV: primary tumor any stage, regional lymph node any stage, distant metastasis present.
  Participants
    Stage III B | 44 | 47 | 91
    Stage IV | 420 | 415 | 835

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Patients Treated With Carboplatin, Paclitaxel and Sorafenib to OS in Patients Treated With Carboplatin, Paclitaxel and Placebo
Description: Overall survival determined as the time (days) from the date of randomization at start of study to the date of death, due to any cause. Outcome measure was assessed regularly, i.e. every 3 weeks during study treatment and every 3 months during post-treatment.
Time Frame: Outcome measure was assessed every 3 weeks starting from randomization, during treatment period and every 3 months during follow-up period until death was recorded or up to data cutoff (1Oct2007) used for planned formal interim analysis
Population: Evaluations of OS based on the ITT population. Subjects alive at the time of analysis were censored at their last date of follow-up (last visit or contact or at the data cut-off date). In the case of an incomplete date, if the day is missing, day 15 (the middle of the month) will be used.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib + C/P | Placebo + C/P
Number analyzed (Participants) | 464 | 462
days | 324 [277 to 423] | 322 [293 to 366]
Statistical Analysis 1: Comparison: Sorafenib + C/P vs Placebo + C/P; Sample size based on primary efficacy endpoint of OS. Clinically meaningful improvement defined as 30% improvement in median OS (i.e. HR of 0.76923, Sorafenib+C/P over Placebo+C/P -Null: theta>=1, Alternative: theta<=0.76923). With overall one-sided alpha of 0.025, 90% power and randomization of 1:1, one formal interim analysis and one final analysis were planned using O'Brien-Fleming type error spending function, and a total of 614 events (deaths) were required; Test type: Superiority or Other; p = 0.915, Log Rank — According to protocol specified O'Brien-Fleming type alpha spending function and 384 deaths at interim analysis (IA), one-sided alpha value for IA was 0.0046; Hazard Ratio (HR) = 1.15, 95% CI [0.94 to 1.41] — Two treatment groups compared using one-sided log-rank test (Sorafenib+C/P over Placebo+C/P) with overall alpha of 0.025 stratified by same stratification factors as randomization

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS determined as time (days) from the date of randomization at start of study to disease progression (radiological or clinical) or death due to any cause, if death occurs before progression.
Time Frame: Tumor measurements and assessments based on RECIST criteria were performed every 6 weeks for the first 18 weeks of therapy ( week 6, 12, and 18) and every 12 weeks thereafter up to data cutoff (1Oct2007) used for planned formal interim analysis
Population: PFS (based on the ITT population) for subjects without disease progression/death at the time of analysis were censored at the last evaluation date. PFS for surviving subjects without post-baseline tumor assessments were censored at one day. In the case of an incomplete date (missing day), day 15 (the middle of the month) will be used.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib + C/P | Placebo + C/P
Number analyzed (Participants) | 464 | 462
days | 139 [132 to 160] | 163 [134 to 175]
Statistical Analysis 1: Comparison: Sorafenib + C/P vs Placebo + C/P; Two treatment groups compared using one-sided log-rank test (Sorafenib+C/P over Placebo+C/P) with alpha of 0.025 stratified by same stratification factors at randomization; Test type: Superiority or Other; p = 0.433, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI [0.84 to 1.16]

3. Secondary Outcome: Overall Best Response
Description: Best overall tumor response for the ITT population was determined according to Response Evaluation Criteria in Solid Tumors (RECIST). Categories: complete response (CR, tumor disappears), partial response (PR, sum of lesion sizes decreased), stable disease (SD, steady state of disease), progressive disease (PD, sum of lesion sizes increased).
Time Frame: as for outcome 2
Population: Evaluations of overall best response rate based on the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib + C/P | Placebo + C/P
Number analyzed (Participants) | 464 | 462
percentage of participants
  Complete Response (CR) | 0.0 | 1.1
  Partial Response (PR) | 27.4 | 22.9
  Stable Disease (SD) | 45.9 | 47.8
  Progressive Disease (PD) | 9.9 | 17.5
  Not evaluated | 16.8 | 10.6
  Disease control | 49.8 | 56.3
Statistical Analysis 1: Comparison: Sorafenib + C/P vs Placebo + C/P; Objective response rate (ie. CR+PR rate) was compared between treatment arms using Cochran-Mantel-Haenszel test with one-side alpha 0.025 adjusting for same stratification factors as randomization; Test type: Superiority or Other; p = 0.1015, Cochran-Mantel-Haenszel — no adjustments; difference in response rate (CR+PR rate) = -3.65, 95% CI [-9.18 to 1.89] — difference in response rates (Complete Response (CR) + Partial Response (PR)) = Placebo+C/P - Sorafenib+C/P

4. Secondary Outcome: Duration of Response
Description: Duration of response (PR or better) is defined as the time from the first documented objective response of PR or CR, whichever is noted earlier, to disease progression or death (if death occurs before progression is documented).
Time Frame: as for outcome 2
Population: Evaluations of duration of response based on the ITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib + C/P | Placebo + C/P
Number analyzed (Participants) | 127 | 111
days | 168 [142 to 184] | 134 [126 to 165]

5. Secondary Outcome: Patient Reported Outcome as Assessed by FACT-L Score. Change From Baseline in Total FACT-L at Cycles 3,5,7,9 and End of Treatment (EOT)
Description: Functional Assessment of Cancer Therapy - Lung cancer subscore (FACT-L). Patient reported outcome as assessed by FACT-L score. FACT-L questionnaire comprises statements about physical, social / family, emotional and functional well-being as well as additional concerns which have to be rated by the patients (0="not at all" to 4="very much"). Cycle duration defined as 21 days. Change from baseline in Total FACT-L on day 1 of cycles 3,5,7,9 (weeks 7,13,19 and 25) and end of treatment (EOT); cycle 1, day 1 used as baseline. EOT is determined by patient's last visit after treatment discontinuation.
Time Frame: Outcome measure was assessed on Day 1 of Cycle 1 and Day 1 of every other cycle (i.e. Cycle 3, 5, 7 etc.) during treatment and at end of treatment visit or up to data cutoff (10ct2007) used for planned formal interim analysis
Population: Evaluations of Total FACT-L based on the ITT population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib + C/P | Placebo + C/P
Number analyzed (Participants) | 464 | 462
Scores on a scale
  Cycle 3, Day 1 | 0.0 (8.0) | 0.1 (9.7)
  Cycle 5, Day 1 | -1.4 (10.5) | -1.3 (9.8)
  Cycle 7, Day 1 | -0.8 (8.1) | -0.5 (9.4)
  Cycle 9, Day 1 | -1.2 (8.0) | -0.6 (10.6)
  End of treatment (EOT) | -3.1 (10.6) | -2.7 (10.5)

6. Secondary Outcome: Patient Reported Outcome as Assessed by LCS Subscale Score. Change From Baseline in LCS Subscale at Cycles 2 Through 9 and at End of Treatment (EOT)
Description: Lung Cancer Symptoms (LCS) subscale ranges from 0 (severe debilitation) to 28 (asymptomatic). Cycle duration defined as 21 days. Change from baseline in LCS Subscale on day 1 of cycles 2 through 9 (weeks 4,7,10,13,16,19,22 and 25) and end of treatment (EOT); cycle 1, day 1 used as baseline. EOT is determined by patient's last visit after treatment discontinuation.
Time Frame: Outcome measure was assessed on Day 1 of Cycle 1 and Day 1 of every cycle (i.e. Cycle 2, 3, 4, 5 etc.) during treatment and at end of treatment visit or up to data cutoff (10ct2007) used for planned formal interim analysis
Population: Evaluations of LCS Subscale based on the ITT population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib + C/P | Placebo + C/P
Number analyzed (Participants) | 464 | 462
Scores on a scale
  Cycle 2, Day 1 | 0.0 (2.7) | -0.1 (3.1)
  Cycle 3, Day 1 | -0.4 (2.9) | -0.2 (2.9)
  Cycle 4, Day 1 | -0.6 (2.9) | -0.3 (3.0)
  Cycle 5, Day 1 | -0.6 (2.9) | -0.5 (2.9)
  Cycle 6, Day 1 | -0.8 (2.9) | -0.4 (3.1)
  Cycle 7, Day 1 | -0.8 (3.1) | -0.4 (2.9)
  Cycle 8, Day 1 | -1.2 (3.2) | -0.2 (2.6)
  Cycle 9, Day 1 | -0.9 (3.1) | -0.3 (3.3)
  End of treatment (EOT) | -0.9 (3.2) | -0.4 (3.0)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from the first subject's first visit (13 Feb 2006) to the planned formal interim analysis (01 Oct 2007 data cut-off date), and additional safety data were collected until the last subject's last visit (05 Feb 2009).
Arm/Group | Sorafenib + C/P | Placebo + C/P
Serious Adverse Events (participants affected / at risk) | 272/463 | 195/459
Other Adverse Events (participants affected / at risk) | 454/463 | 450/459
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + C/P (N=463) | Placebo + C/P (N=459)
Allergic reaction (Immune system disorders) | 11 | 4
Neutrophils (Blood and lymphatic system disorders) | 15 | 7
Hemoglobin (Blood and lymphatic system disorders) | 11 | 8
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Platelets (Blood and lymphatic system disorders) | 8 | 2
Leukocytes (Blood and lymphatic system disorders) | 2 | 1
Supraventricular arrhythmia, atrial fibrillation (Cardiac disorders) | 2 | 1
Conduction abnormality, asystole (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia, sinus bradycardia (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia, supravent extrasystoles (pac;premnodal/junct contr) (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia, supraventricular tachycardia (Cardiac disorders) | 3 | 0
Supraventricular arrhythmia, sinus tachycardia (Cardiac disorders) | 2 | 0
vasovagal episode (Cardiac disorders) | 0 | 1
Ventricular arrhythmia, ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular arrhythmia, ventricular arrhythmia NOS (Cardiac disorders) | 0 | 1
Ventricular arrhythmia, ventricular tachycardia (Cardiac disorders) | 0 | 1
Cardiopulmonary arrest (Cardiac disorders) | 3 | 2
Pericardial effusion (Cardiac disorders) | 0 | 3
Hypertension (Cardiac disorders) | 2 | 2
Cardiac ischemia/infarction (Cardiac disorders) | 3 | 4
Hypotension (Cardiac disorders) | 1 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Death not associated with CTCAE term, death NOS (General disorders) | 4 | 2
Death not associated with CTCAE term, disease progression NOS (General disorders) | 23 | 24
Death not associated with CTCAE term, multi-organ failure (General disorders) | 0 | 1
Death not associated with CTCAE term, sudden death (General disorders) | 3 | 1
Diabetes (Endocrine disorders) | 1 | 0
Fever (General disorders) | 17 | 10
Fatigue (General disorders) | 5 | 4
Weight loss (General disorders) | 1 | 0
Constitutional symptoms - other (General disorders) | 19 | 13
Rigors/chills (General disorders) | 1 | 0
Anorexia (Gastrointestinal disorders) | 3 | 2
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Dehydration (Gastrointestinal disorders) | 9 | 4
Diarrhea (Gastrointestinal disorders) | 5 | 6
Dysphagia (Gastrointestinal disorders) | 1 | 2
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Mucositis (clinical exam), oral cavity (Gastrointestinal disorders) | 1 | 0
Necrosis, GI, anus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 5
Ileus (Gastrointestinal disorders) | 2 | 2
Perforation, GI, colon (Gastrointestinal disorders) | 1 | 0
Ulcer, GI, stomach (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2
Hemorrhage, GI, abdomen NOS (Vascular disorders) | 2 | 0
Hemorrhage, GI, colon (Vascular disorders) | 0 | 2
Hemorrhage, GI, duodenum (Vascular disorders) | 1 | 0
Hemorrhage, GI, stomach (Vascular disorders) | 0 | 1
Hemorrhage, GI, lower GI NOS (Vascular disorders) | 1 | 0
Hemorrhage, GI, upper GI, NOS (Vascular disorders) | 0 | 1
Hemorrhage pulmonary, bronchopulmonary NOS (Vascular disorders) | 0 | 2
Hemorrhage pulmonary, bronchus (Vascular disorders) | 0 | 1
Hemorrhage pulmonary, lung (Vascular disorders) | 11 | 8
Hemorrhage pulmonary, nose (Vascular disorders) | 1 | 0
Hemorrhage pulmonary, respiratory tract NOS (Vascular disorders) | 5 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Hepatobilary - other (Hepatobiliary disorders) | 0 | 1
Pancreatitis (Hepatobiliary disorders) | 1 | 0
Infection (documented clinically), abdomen NOS (Infections and infestations) | 1 | 0
Infection (documented clinically), blood (Infections and infestations) | 9 | 0
Infection (documented clinically), bladder (urinary) (Infections and infestations) | 0 | 1
Infection (documented clinically), bronchus (Infections and infestations) | 1 | 3
Infection (documented clinically), lung (pneumonia) (Infections and infestations) | 25 | 10
Infection (documented clinically), pleura (empyema) (Infections and infestations) | 0 | 1
Infection (documented clinically), skin (cellulitis) (Infections and infestations) | 2 | 0
Infection (documented clinically), upper airway NOS (Infections and infestations) | 2 | 1
Infection (documented clinically), urinary tract NOS (Infections and infestations) | 1 | 0
Infection (documented clinically), vein (Infections and infestations) | 0 | 1
Infection with normal ANC, blood (Infections and infestations) | 2 | 2
Infection with normal ANC, bronchus (Infections and infestations) | 1 | 3
Infection with normal ANC, catheter-related (Infections and infestations) | 1 | 0
Infection with normal ANC, colon (Infections and infestations) | 0 | 1
Febrile neutropenia (Infections and infestations) | 16 | 8
Infection with normal ANC, lung (pneumonia) (Infections and infestations) | 6 | 3
Infection with normal ANC, upper airway NOS (Infections and infestations) | 1 | 0
Infection - other (Infections and infestations) | 2 | 1
Infection with unknown ANC, anal/perianal (Infections and infestations) | 0 | 1
Infection with unknown ANC, lung (pneumonia) (Infections and infestations) | 5 | 2
Infection with unknown ANC, pleura (empyema) (Infections and infestations) | 0 | 1
Edema: limb (Blood and lymphatic system disorders) | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 2 | 6
Muscuskeletal - other (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness, extremity-lower (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle weakness, whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 | 1
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 | 0
ALT (Metabolism and nutrition disorders) | 2 | 0
AST (Metabolism and nutrition disorders) | 1 | 0
Creatinine (Metabolism and nutrition disorders) | 1 | 0
GGT (Metabolism and nutrition disorders) | 1 | 0
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Mood alteration, agitation (Nervous system disorders) | 1 | 0
CNS ischemia (Nervous system disorders) | 1 | 7
Confusion (Nervous system disorders) | 6 | 3
Dizziness (Nervous system disorders) | 3 | 2
Mood alteration, euphoria (Nervous system disorders) | 0 | 1
Speech impairment (Nervous system disorders) | 1 | 0
Mood alteration, depression (Nervous system disorders) | 3 | 0
Neuropathy: motor (Nervous system disorders) | 1 | 1
Neurology - other (Nervous system disorders) | 2 | 5
Neuropathy: sensory (Nervous system disorders) | 3 | 6
Seizure (Nervous system disorders) | 3 | 1
Somnolence (Nervous system disorders) | 2 | 0
Syncope (fainting) (Nervous system disorders) | 1 | 1
Pain, back (General disorders) | 4 | 2
Pain, chest/thorax NOS (General disorders) | 0 | 5
Pain, chest wall (General disorders) | 1 | 1
Pain, tumor pain (General disorders) | 2 | 4
Pain, abdomen NOS (General disorders) | 3 | 2
Pain, joint (General disorders) | 2 | 0
Pain, muscle (General disorders) | 0 | 1
Pain, bone (General disorders) | 3 | 1
Pain, liver (General disorders) | 1 | 0
Pain, pain NOS (General disorders) | 1 | 0
Pain, stomach (General disorders) | 1 | 0
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Fistula, pulmonary, bronchus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fistula, pulmonary, lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Airway obstruction, bronchus (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 17 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 24 | 23
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cystitis (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 4 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 | 0
Intraop injury, bone (Injury, poisoning and procedural complications) | 1 | 0
Syndromes - other (General disorders) | 1 | 0
Thrombosis/embolism (vascular access) (Vascular disorders) | 0 | 3
Vascular - other (Vascular disorders) | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 16 | 17
Bone marrow cellularity (Blood and lymphatic system disorders) | 1 | 2
Supraventricular arrhythmia, atrial (Cardiac disorders) | 1 | 0
cardiac general - other (Cardiac disorders) | 1 | 1
ascites (Gastrointestinal disorders) | 1 | 0
Fistula, GI, abdomen NOS (Gastrointestinal disorders) | 0 | 1
perforation, GI, stomach (Gastrointestinal disorders) | 1 | 0
Hematoma (Blood and lymphatic system disorders) | 0 | 1
Hemorrhage, GI, esophagus (Blood and lymphatic system disorders) | 0 | 1
Hemorrhage, Gu, bladder (Blood and lymphatic system disorders) | 1 | 0
Infection (documented clinically), anal/perianal (Infections and infestations) | 1 | 0
Infection (documented clinically), mucosa (Infections and infestations) | 1 | 0
Infection with normal ANC, anal/perianal (Infections and infestations) | 2 | 0
Infection with normal ANC, pleura (empyema) (Infections and infestations) | 1 | 0
Infection with normal ANC, urethra (Infections and infestations) | 1 | 0
Opportunistic infection (Infections and infestations) | 1 | 0
Infection with unknown ANC, blood (Infections and infestations) | 0 | 2
Infection with unknown ANC, muscle (infection myositis) (Infections and infestations) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Pain, neck (General disorders) | 1 | 0
Bruising (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Skin and subcutaneous tissue disorders) | 1 | 0
Intraop injury, lung (Surgical and medical procedures) | 1 | 0
Flu-like syndrome (General disorders) | 1 | 0
Peripheral arterial ischemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + C/P (N=463) | Placebo + C/P (N=459)
Neutrophils (Blood and lymphatic system disorders) | 170 | 168
Hemoglobin (Blood and lymphatic system disorders) | 145 | 148
Platelets (Blood and lymphatic system disorders) | 140 | 67
Leukocytes (Blood and lymphatic system disorders) | 78 | 67
Hypertension (Cardiac disorders) | 90 | 46
Fever (General disorders) | 85 | 60
Insomnia (General disorders) | 79 | 83
Fatigue (General disorders) | 251 | 228
Weight loss (General disorders) | 99 | 57
Anorexia (Gastrointestinal disorders) | 149 | 122
Constipation (Gastrointestinal disorders) | 126 | 107
Diarrhea (Gastrointestinal disorders) | 205 | 107
Heartburn (Gastrointestinal disorders) | 47 | 26
Mucositis (clinical exam), oral cavity (Gastrointestinal disorders) | 77 | 33
Nausea (Gastrointestinal disorders) | 201 | 204
Vomiting (Gastrointestinal disorders) | 122 | 108
Edema: limb (Blood and lymphatic system disorders) | 52 | 51
Dizziness (Nervous system disorders) | 55 | 52
Neuropathy: sensory (Nervous system disorders) | 236 | 250
Pain, back (General disorders) | 50 | 53
Pain, chest/thorax NOS (General disorders) | 70 | 70
Pain, extremity-limb (General disorders) | 69 | 58
Pain, abdomen NOS (General disorders) | 60 | 50
Pain, head/headache (General disorders) | 52 | 50
Pain, joint (General disorders) | 83 | 100
Pain, muscle (General disorders) | 96 | 120
Pain, bone (General disorders) | 52 | 41
Cough (Respiratory, thoracic and mediastinal disorders) | 142 | 138
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 138 | 136
Alopecia (Skin and subcutaneous tissue disorders) | 214 | 215
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 113 | 24
Pruritus (Skin and subcutaneous tissue disorders) | 66 | 35
Rash/desquamation (Skin and subcutaneous tissue disorders) | 239 | 80
Allergic reaction (Immune system disorders) | 29 | 30
Hypotension (Cardiac disorders) | 36 | 28
Sweating (General disorders) | 30 | 31
Dehydration (Gastrointestinal disorders) | 36 | 16
Mucositis (functional/symptomatic), oral cavity (Gastrointestinal disorders) | 25 | 12
Taste alteration (Gastrointestinal disorders) | 43 | 38
Hemorrhage pulmonary, nose (Vascular disorders) | 46 | 21
Pain, throat / pharynx / larynx (General disorders) | 24 | 17
Hypokalemia (Metabolism and nutrition disorders) | 46 | 25
Hypomagnesemia (Metabolism and nutrition disorders) | 40 | 26
Mood alteration, anxiety (Nervous system disorders) | 42 | 35
Mood alteration, depression (Nervous system disorders) | 28 | 20
Voice changes (Respiratory, thoracic and mediastinal disorders) | 28 | 22
Dry skin (Skin and subcutaneous tissue disorders) | 41 | 24
Erythema multiforme (Skin and subcutaneous tissue disorders) | 25 | 4
Pain, tumor pain (General disorders) | 22 | 23
Rhinitis (Immune system disorders) | 18 | 23
Muscle weakness, whole body / generalized (Musculoskeletal and connective tissue disorders) | 27 | 20
Hyperglycemia (Metabolism and nutrition disorders) | 19 | 23

LIMITATIONS AND CAVEATS:
Based on the results of the interim analysis, it was determined that the study would not meet its primary efficacy endpoint and the study was terminated early. The planned biomarker analysis was suspended due to early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less